CLINICAL TRIAL: NCT05066503
Title: Nutritional Therapy for Delirium in Elderly Hospitalized Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 260279
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Subacute Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delirious subjects receiving active study product (Active Comparator): Subjects will ingest an oral amino-acid containing nutritional supplement twice daily for up to 4 days.
  Interventions: Dietary Supplement: 260279 active study product
- Control group (No Intervention): Delirious control group and non-delirious control group who receives standard treatment in the hospital.

INTERVENTIONS:
Dietary Supplement: 260279 active study product — The active study product (20g per serving) contains 13.6g of amino acids and natural flavors, citric acid, malic acid, and stevia for flavoring.
  Other Names: there is not a non-proprietary name for this supplement.
  Arms: Delirious subjects receiving active study product

SUMMARY:
The investigators have developed a proprietary blend of amino acids that they think will help to prevent or reduce the severity of delirium in older adults (60 years and older) who are hospitalized for certain infections. In this study, up to 60 people will be enrolled.20 will be asked to drink this blend twice a day for up to 4 days, and 20 will receive standard treatment in the hospital for the same time period. The other 20 subjects will be non-delirious control subjects who do not consume any study products.

DETAILED DESCRIPTION:
This will be an interventional pilot study to determine the effectiveness of a specific amino acid supplement developed by the investigators versus standard treatment in mitigating delirium in geriatric patients hospitalized at UAMS for certain infections. Up to 40 delirious and 20 non-delirious subjects (Aged 60 years and older) of any gender or ethnicity will be enrolled (60 subjects maximum). Twenty patients with delirium will be asked to drink this blend twice a day for up to 4 days, and 20 patients with delirium will receive standard treatment in the hospital for the same time period. The other 20 subjects will be non-delirious control subjects who do not consume any study products. All subjects will undergo 2-5 blood draws and 3-7 cognitive assessments while they are admitted to the hospital, depending on study group assignment and discharge date.

ELIGIBILITY:
Inclusion Criteria: Delirious cohort

1. Aged 60 years and older.
2. Documented presence of either delirium, acute confusion, or altered mental status in medical record.
3. Currently hospitalized with a diagnosis of one of the following:

   1. sepsis/septicemia
   2. Pneumonia
   3. Urinary tract infection
   4. Clostridium-difficile infection
   5. Other bone or tissue infection
   6. Fever of unknown origin

Inclusion Criteria: NON-Delirious cohort

1. Aged 60 years and older.
2. Current diagnosis of one of the following:

   1. sepsis/septicemia
   2. Pneumonia
   3. Urinary tract infection
   4. Clostridium-difficile infection
   5. Other bone or tissue infection
   6. Fever of unknown origin

Exclusion Criteria: all subjects

1. Chronic kidney disease (eGFR <30).
2. Admitted to the hospital for major psychiatric illness.
3. Major psychiatric illness not controlled by medication/treatment.
4. Delirium etiology of drug overdose or alcohol withdrawal.
5. Major surgery within the past five days.
6. Known or suspected Covid-19 positive.
7. Continuous feeding tube

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in CAM-S (Confusion Assessment Method-Short) and 4 AT score from baseline to day 3 or up to day 4. | As determined over an up to 4-day intervention duration.
  CAM-S and 4 AT is a tool to determine and quantify delirium. Subjects in the non-control arms will undergo this test twice each day. The score ranges from 0-7, with lower numbers being better (little to no signs of delirium).

CONTACTS AND LOCATIONS:
Overall Officials: Gohar Azhar, M.D., Principal Investigator — University of Arkansas
Locations (1):
- UAMS Center on Aging, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No